CLINICAL TRIAL: NCT01722435
Title: Completion of Substitution Treatment With Methadone/Levomethadone - a Prospective Study
Brief Title: Completion of OST - a Prospective Study
Status: Completed | Type: Observational
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Collaborators: Asklepios Kliniken Hamburg GmbH (Other); Dr. Rainer Ullmann (Unknown); Dr. Sibylle Quellhorst (Unknown); Dr. Jochen Brack (Unknown); Michael Klemperer (Unknown); Gesine Hoeft (Unknown)
Responsible Party: Principal Investigator, Prof. Dr. med. Jens Reimer, Prof. Dr., Universitätsklinikum Hamburg-Eppendorf
Other Study IDs: ZIS-OST-PV3718
Record Dates: First submitted 2012-11-02; First posted 2012-11-06 (Estimated); Results first posted 2014-08-22 (Estimated); Last update posted 2019-10-09 (Actual); Status verified 2019-10

CONDITIONS: Opioid Dependence
Keywords: opioid dependence; opiate substitution treatment; methadone; completion; termination
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Opiate Substitution Treatment

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- OST completers: Patients who are likely to complete OST during the next 12 or 18 months
  Interventions: Drug: Opiate Substitution Treatment

INTERVENTIONS:
Drug: Opiate Substitution Treatment

SUMMARY:
Only limited information on the process of completing long-term opiate substitution treatment (OST) with substances like methadone exist. Furthermore, systematic knowledge from scientific studies is scarce, there are only few studies with respect to treatment completion or regular termination (mainly catamnestic analyses). Studies by Nordt et al. (2004) or Nordt & Stohler (2006) show an estimated rate of 10% of patients per year who terminate OST by means of tapering the substitution agent or changing into withdrawal treatment in specialized clinics. It is state of the art that an indication for termination of OST has to be based on a common agreement between the patient and the doctor. Furthermore, the patient should live in a stable social situation and the state of health had markedly improved. Finally, the patient has to be free of (illegal) drug use for at least 6 months and the individual aims of treatment should have been reached (Vader et al. 2003).

The main objective of the prospective and explorative study is the systematic description of the process of termination of OST. With a comparison between patients who complete OST regularly and patients who terminate treatment prematurely (or are still in treatment) predictors of positive termination of OST can be identified.

Patients treated with methadone or levomethadone of 5 general practitioners' practices and 2 specialized clinics who might be able to terminate OST during the next 12 months from the doctors' perspective can take part in the study. In addition to baseline examination further assessments take place every 3 months (i.e. after 3, 6, 9 and 12 months). The questionnaires include state of health, well-being, social situation as well as drug and alcohol use. Furthermore, the treating doctors are asked every 3 months to fill out questionnaires on infections and other disorders, clinical characteristics, dosage process and drug use (measured by urine samples).

Patients who will be successful in completing OST during the observational period will be compared with the remaining cases.

Finally, a 6-month follow-up is planned in order to investigate the stability and maintenance of the situation at month 12.

ELIGIBILITY:
Inclusion Criteria:

* opioid dependence according ICD-10
* Minimum age of 18 years
* In OST with methadone or levomethadone
* Expected or planned treatment completion during the next 12 months
* Informed consent to participate in the study

Exclusion Criteria:

* Patients with planned hospitalisation during the next 12 months
* Patients who are likely or it is save to assume that they will be incarcerated or imprisoned during the next 12 months
* Disability to take part in the study or follow the study conditions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in primary care setting (GPs) or specialized clinics likely to complete opiate substitution treatment (OST) during the next 12 months.
Sampling Method: Non-Probability Sample
Enrollment: 78 (Actual)
Dates: Start 2011-07; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jens Reimer, Professor, Principal Investigator — Centre for Interdisciplinary Addiction Research of Hamburg University

RESULTS

PARTICIPANT FLOW:
Groups:
- OST Completers: Patients who are likely to complete OST during the next 12 or 18 months
  Opiate Substitution Treatment
Period: Overall Study
Arm/Group | OST Completers
Started | 78
Completed | 78
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Patients treated with methadone or levomethadone who were eligible for the study and consented to participate and qualified for treatment completion in the next 12 months.
Groups:
- OST Completers: The main objective of this prospective study was the description of the process of termination of opiate substitution treatment (OST). Patients in primary care setting (GPs) or specialized clinics likely to complete OST during the next 12 months were asked to fill out questionnaires every 3 months over a 12-months period and were followed up another 6 months later. Accordingly, the doctors documented their patients' state of health and provided an evaluation of their living situation every 3 months and at the end of treatment (or - if patients stayed in treatment - at the end of the 18-months study period).
  At the beginning of the study overall 1367 OST patients were treated in the 7 participating clinics and practices. 972 of them were treated with methadone or levomethadone. In line with the inclusion criteria, 97 patients were eligible for the study, 78 of them consented to participate in the study (8.0% of all patients treated with methadone or levomethadone).
Arm/Group | OST Completers
Number analyzed (Participants) | 78
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.5 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54
  Male | 24
Lengths of OST before study entry [Mean (Standard Deviation); unit: months] | 92.9 (59.5)
Participants on specific medication [Number; unit: participants]
  d,l-methadone | 37
  levometahdone | 37
  buprenorphine | 4
Average dose of medication taken [Mean (Standard Deviation); unit: milligrams]
  d,l-methadone | 54.8 (41.8)
  levomethadone | 26.6 (21.6)
  buprenorphine | 14.3 (8.2)

OUTCOME MEASURES:

1. Primary Outcome: Completion of OST
Description: Regularly completion of OST, i.e. not being on opioid medication any more, during the study period.
Time Frame: 18 months
Measure: Number; unit: participants
Arm/Group | OST Completers
Number analyzed (Participants) | 78
participants | 9

2. Primary Outcome: OST Drop-outs
Description: Participants dropped out of OST Treatment during the study period.
Time Frame: 18 months
Measure: Number; unit: participants
Arm/Group | OST Completers
Number analyzed (Participants) | 78
participants | 15

3. Secondary Outcome: Mean Time to Complete OST
Description: Mean time of study participation (M, SD) until Treatment completion or end of study (after 18 months).
Time Frame: 18 months
Measure: Mean (Standard Deviation); unit: days
Groups:
- OST Completers: Patients completed OST during 12 or 18 months.
Arm/Group | OST Completers
Number analyzed (Participants) | 9
days | 232 (159)

4. Secondary Outcome: Mean Time to Drop-out of OST
Description: Mean time of study participation (M, SD) until drop-out of treatment.
Time Frame: 18 months
Measure: Mean (Standard Deviation); unit: days
Groups:
- OST Drop-outs: Patients dropped out of OST during 12 or 18 months.
Arm/Group | OST Drop-outs
Number analyzed (Participants) | 15
days | 315 (195)

5. Secondary Outcome: Mean Time Staying in OST
Description: Mean time of study participation (M, SD) of patients who stayed in OST Treatment until end of study (after 18 months).
Time Frame: 18 months
Measure: Mean (Standard Deviation); unit: days
Groups:
- Still in OST Completers: Patients still in OST during the whole study period.
Arm/Group | Still in OST Completers
Number analyzed (Participants) | 54
days | 549 (91)

ADVERSE EVENTS:
Arm/Group | OST Completers
Serious Adverse Events (participants affected / at risk) | 0/78
Other Adverse Events (participants affected / at risk) | 0/78

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No